CLINICAL TRIAL: NCT05485376
Title: The Pulmonary Artery Catheter in Cardiogenic Shock Trial
Brief Title: Pulmonary Artery Catheter in Cardiogenic Shock Trial
Acronym: PACCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00002564
Record Dates: First submitted 2022-06-17; First posted 2022-08-03 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Cardiogenic Shock; Heart Failure
Keywords: Pulmonary Artery Catheter
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Pulmonary Artery Catheter (Experimental): If you are in the experimental group a PAC will be placed within 6 hours of randomization and within 24 hours of presentation with ADHF-CS.
  Interventions: Device: Pulmonary Artery Catheter
- No or delayed Pulmonary Artery Catheter (No Intervention): If you are in the control group, a PAC will not be placed during hospitalization or may be placed 48 hours after randomization into the study. Placement of a PAC within 48 hours is only permitted for emergencies.

INTERVENTIONS:
Device: Pulmonary Artery Catheter — The pulmonary artery catheter (PAC) is a diagnostic instrument that enables continuous hemodynamic monitoring of cardiac filling pressures, cardiac output, and pulmonary pressures.
  Arms: Early Pulmonary Artery Catheter

SUMMARY:
The primary objective of the PACCS trial is to assess if early invasive hemodynamic assessment and ongoing management with a PAC in patients with cardiogenic shock due to acutely decompensated heart failure (AHDF-CS) is associated with lower in-hospital mortality risk compared to the current standard of care with no or delayed PAC assessment.

DETAILED DESCRIPTION:
The PACCS trial is a multicenter, randomized, parallel group, adaptive trial that will test the hypothesis that early invasive hemodynamic assessment (within 6 hours of randomization) and ongoing management with a PAC decreases in-hospital mortality compared to clinical management with delayed (beyond 48 hours after randomization) or no PAC-guided assessment among patients with cardiogenic shock due to acutely decompensated heart failure (AHDF-CS). The trial uses an adaptive sample size re-estimation design. An interim analysis will be performed when the primary endpoint is available for 200 participants and may lead to an increase in the target sample size (minimum sample size 400, maximum sample size 800).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤90 years
2. Clinical heart failure presentation and left ventricular function as follows: Either 2A or 2B must be present A. Subject has de novo acute decompensated heart failure and shock with an LVEF ≤40% OR B. Subject has acute on chronic heart failure with a documented history of a LVEF ≤40% within 6 months of admission and a current LVEF ≤40% within 24 hours of screening during the current hospitalization.

   NOTE: The LVEF must be quantitatively measured as ≤ 40% by an echocardiogram within 24 hours of screening. If multiple echocardiograms have been performed within 24 hours, the most recent test must be used to qualify the patient.
3. Cardiogenic Shock (CS) defined by a lactate level ≥ 2.1 mmol/L and any 2 of the following parameters within 24 hours of screening:

   1. SBP <90 mmHg for more than 30 minutes from baseline SBP
   2. Requires the use of at least 1 vasopressor or inotrope
   3. Requires intra-aortic balloon pump (IABP) support
   4. Presence of congestion on exam: JVP elevated, pulmonary edema on CXR or exam, dyspnea at rest, orthopnea, bendopnea, or worsening peripheral or abdominal swelling
4. Initial diagnosis of CS within 24 hours of screening at the enrolling site
5. Patient or legally authorized representative provides informed consent

A HIPAA waiver for screening is requested to identify potential subjects. No recruitment materials will be given to potential subjects. No identifiable data will be retained for subjects that are determined to be ineligible

Exclusion Criteria:

1. Primary etiology of shock other than systolic left heart failure including but not limited to: acute myocardial infarction, sepsis, hypovolemia, hemorrhage, severe anemia, primary RV failure, pulmonary embolism, or tamponade.
2. Patient has a durable ventricular assist device or temporary mechanical circulatory support (other than IABP) or PAC prior to enrollment
3. Actively listed for cardiac transplantation (Status 7 patients are eligible for the trial)
4. Patient transferred from another facility with a diagnosis of cardiogenic shock
5. Any known co-morbidity other than heart failure with anticipated survival < 6 months
6. Pre-enrollment labs (any of the following): International Normalized Ratio (INR) > 3, Platelet count < 50k, Hemoglobin < 7
7. Refractory or recurrent cardiac arrest (>1 episode requiring defibrillation or cardiopulmonary resuscitation) within 24 hours prior to screening
8. DNR/ DNI status
9. Pregnancy, child-birth within 6 months, or lactation
10. Active infection documented by persistent fever (Temp > 38.4oC within 24 hours of screening) or confirmed bacteremia
11. Implantation of PPM or ICD within past 3 months
12. Mechanical complication of AMI (ie VSD, papillary muscle rupture, flail mitral regurgitation, free wall rupture)
13. Anoxic brain injury
14. On renal replacement therapy prior to enrollment
15. Cardiac surgery within 3 months of current admission
16. Severe aortic, pulmonic, tricuspid stenosis or acute structural mitral regurgitation or infective endocarditis
17. History of cardiac amyloid
18. Congenital heart disease excluding the presence of a bicuspid aortic valve
19. Planned cardiac surgery during admission
20. World Health Organization (WHO) Group I, III, IV, or V pulmonary hypertension
21. Any known contraindication to PAC placement
22. Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device that has not reached its primary endpoint
23. Any medical or psychiatric condition such as dementia, alcoholism, or substance abuse which may preclude informed consent or interfere with any of the study procedures, including follow-up
24. Prior stroke with any permanent neurologic deficit or any prior intracranial hemorrhage or any prior subdural hematoma or known intracranial pathology pre-disposing to intracranial bleeding, such as an arteriovenous malformation or mass
25. Subject has previously hospitalized for COVID-19 unless he/she has been discharged and asymptomatic for ≥4 weeks
26. Subject is COVID-19 PCR/antigen positive within the prior 4 weeks
27. Subject belongs to a vulnerable population [defined as individuals with mental disability, persons in nursing homes, impoverished persons, homeless persons, nomads, refugees and those permanently incapable of giving informed consent; vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, members of the armed forces and persons kept in detention]

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who die in the hospital | Length of stay in hospital, an average of 30 days

SECONDARY OUTCOMES:
Number of Participants with in-hospital Cardiac Arrest | Length of stay in hospital, an average of 30 days
Number of Participants that require Mechanical Ventilation | Length of stay in hospital, an average of 30 days
Number of Participants that require Renal Replacement Therapy | Within 96 hours of randomization
Length of stay in CCU or ICU | Length of stay in hospital, an average of 30 days
Occurrence of heart transplantation and durable LVAD implantation | Length of stay in hospital, an average of 30 days
Death | 30 days and 6 months after discharge
Heart failure hospitalizations/emergency room visits | 30 days and 6 months after discharge
Admission to an outpatient IV diuretic center | 30 days and 6 months after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Navin K Kapur, MD, Principal Investigator — nkapur@tuftsmedicalcenter.org
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Filipescu R, Collins SP, Radu RI, Ben Gal T, Antohi L, Abdelhamid M, Geavlete O, Pana M, Farmakis D, Matei DC, Savarese G, Margineanu C, Polovina M, Miro O, Guz D, Palazzuoli A, Masip J, Adamo M, Ambrosy AP, Chioncel O. Therapeutic Advances in the Management of Cardiogenic Shock. Am J Ther. 2026 Jan 15. doi: 10.1097/MJT.0000000000002025. Online ahead of print. PMID 41543923